CLINICAL TRIAL: NCT03604549
Title: Therapeutic Effect of Sonographic Hysterosalpingography: Oil vs Water Based Media
Brief Title: Sonographic Hysterosalpingography: Oil vs Water Based Media (SHOW Trial)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Interim Chair and Vice Chair of Research, Department of Obstetrics and Gynecology, Professor of Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00008466
Record Dates: First submitted 2018-07-10; First posted 2018-07-27 (Actual); Results first posted 2022-02-24 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline (Placebo Comparator): Women in this arm will receive a flush with saline after normal saline Sono HSG.
  Interventions: Drug: Saline
- Lipiodol UF (Experimental): Women in this arm will receive a flush with Lipiodol UF after normal saline Sono HSG.
  Interventions: Drug: Lipiodol UF

INTERVENTIONS:
Drug: Lipiodol UF — Up to 10cc of Lipiodol Ultra Fluid will be infused via intrauterine catheter
  Other Names: Lipiodol Ultra Fluid
  Arms: Lipiodol UF
Drug: Saline — Up to 10cc of saline will be infused via intrauterine catheter
  Arms: Saline

SUMMARY:
Performing fluoroscopic HSG with oil based contrast medium has been shown to increase pregnancy rates in a subfertile population. This is a pilot study to test the efficacy of as well as the tolerability and safety of using lipid based oil medium for sonographic based hysterosalpingography (Sono HSG) compared to water based contrast (i.e. normal saline) for women seeking fertility. The double blind study will randomize 56 women at the time of Sono HSG in a 1:1 ratio to receive through the SHG catheter either up to 10 cc of Lipiodol UF® or normal saline. The investigators will collect subjective pain experience and follow the subjects for 6 months after the test for pregnancy and collect all adverse events during and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for Sono HSG for fertility testing
* In good general health
* Willing and capable of complying with the study procedures
* At least one patent tube and no endometrial pathology on Sono HSG
* Ready to undergo infertility treatment immediately after the test
* Not planning on IVF therapy in the next 6 mos

Exclusion Criteria:

* Known tubal or endometrial (polyp, submucous fibroid, etc.) pathology
* At high risk for tubal disease due to history of Pelvic Inflammatory Disease
* Known hypersensitivity to Lipiodol UF®or known allergy to iodine containing contrast media or shellfish
* Endometrial pathology on Sono HSG requiring further evaluation (as per the performing physician)
* Bilateral tubal occlusion on Sono HSG
* Unable to tolerate potential pain associated with the study.
* Requiring IVF due to severe male factor, known pelvic adhesions, etc.
* Couples with decreased male factor fertility rate (i.e., low sperm count or motility, i.e. less than 5 million/mL concentration on semen analysis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Legro, M.D., Principal Investigator — Penn State University and Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang R, Watson A, Johnson N, Cheung K, Fitzgerald C, Mol BWJ, Mohiyiddeen L. Tubal flushing for subfertility. Cochrane Database Syst Rev. 2020 Oct 15;10(10):CD003718. doi: 10.1002/14651858.CD003718.pub5. PMID 33053612

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline: Women in this arm will receive a flush with saline after normal saline Sono Hystersalpingography. .
  Saline: Up to 10cc of saline will be infused via intrauterine catheter
- Lipiodol UF: Women in this arm will receive a flush with Lipiodol UF after normal saline Sono Hystersalpingography.
  Lipiodol UF: Up to 10cc of Lipiodol Ultra Fluid will be infused via intrauterine catheter
Period: Overall Study
Arm/Group | Saline | Lipiodol UF
Started | 29 | 29
Completed | 24 | 24
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Population: Baseline analysis population represents subjects having study agent administered during sono HSG procedure
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Lipiodol UF | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (3.9) | 31.0 (5.4) | 30.3 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 21 | 20 | 41
  Race: Asian | 0 | 2 | 2
  Race: Multi-racial | 3 | 1 | 4
  Race: Unknown | 0 | 1 | 1
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.3 (7.3) | 31.8 (8.9) | 31.0 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Ongoing Pregnancy Rate
Description: 8 week viable intrauterine pregnancy
Time Frame: within 6 months of Sono HSG procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Saline | Lipiodol UF
Number analyzed (Participants) | 24 | 24
Participants | 9 | 4
Statistical Analysis 1: Comparison: Saline vs Lipiodol UF; Test type: Superiority; p = 0.10, Chi-squared; Risk Ratio (RR) = 0.44, 95% CI 2-sided [0.16 to 1.25] — Lipiodol UF is the numerator and Saline is the denominator for RR

2. Secondary Outcome: Procedural Related Pain Assessed by Visual Analog Scale
Description: scale ranges from 0-10 with a higher score indicating more pain
Time Frame: After sono hystersalpingography study infusion/procedure completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline | Lipiodol UF
Number analyzed (Participants) | 24 | 24
units on a scale | 3.5 (2.7) | 3.5 (2.9)
Statistical Analysis 1: Comparison: Saline vs Lipiodol UF; Test type: Superiority; p = 0.96, t-test, 2 sided; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-1.59 to 1.68] — Difference reported as Lipiodol UF - Saline

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Saline | Lipiodol UF
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline (N=24) | Lipiodol UF (N=24)
Cervical ectopic hemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT03604549/Prot_SAP_000.pdf